CLINICAL TRIAL: NCT06354231
Title: A Prospective, Open-label, Single-arm, Clinical Study of Disitamab Vedotin Combined With Toripalimab for Renal Preservation in Solitary Kidney or Renal Insufficiency or Bilateral Multiple Upper Urinary Tract Urothelial Carcinoma
Brief Title: DV Combined With Toripalimab for Renal Preservation in Solitary Kidney or Renal Insufficiency or Bilateral Multiple UTUC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C012
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Renal Insufficiency; Upper Urinary Tract Urothelial Carcinoma; Solitary Kidney
MeSH Terms: conditions — Renal Insufficiency; Solitary Kidney | interventions — toripalimab; Laser Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DV+Toripalimab (Experimental): DV, 2.0 mg/kg, intravenously administered every 2 weeks; toripalimab, 3.0mg/kg, intravenously administered every 2 weeks;
  Interventions: Drug: DV; Drug: Toripalimab; Procedure: Laser surgery

INTERVENTIONS:
Drug: DV — 2.0 mg/kg, intravenously administered every 2 weeks
  Other Names: RC48
Drug: Toripalimab — 3.0mg/kg, intravenously administered every 2 weeks
  Other Names: JS001
Procedure: Laser surgery — Subjects will receive 6 cycles of DV and toripalimab, followed by laser surgery to remove ureteral or renal pelvis tumors, followed by 12 cycles of DV and 1 year of toripalimab consolidation therapy.

SUMMARY:
Approximately 20 participants will be enrolled in the study to evaluate the efficacy and safety of the combination of DV (DV, 2.0 mg/kg, intravenously administered every 2 weeks) and toripalimab (toripalimab, 3.0mg/kg, intravenously administered every 2 weeks). Subjects will receive 6 cycles of DV and toripalimab, followed by laser surgery to remove ureteral or renal pelvis tumors, followed by 12 cycles of DV and 1 year of toripalimab consolidation therapy. Efficacy and safety were evaluated by cystoscopy, ureteroscopy, laboratory tests, and imaging examinations after treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Histologically confirmed isolated renal or renal insufficiency or bilateral upper urinary tract urothelial carcinoma;
* Refusal or ineligibility for RNU;
* Preoperative risk stratification was defined as high-risk UTUC, defined as patients with any of the following factors:

  1. Hydronephrosis;
  2. Tumor diameter ≥2cm;
  3. Urine cytology suggests a high-grade tumor;
  4. A ureteroscopic biopsy suggests a high-grade tumor;
  5. CT showed a localized invasion;
  6. Multifoci diseases;
  7. With multiple histological subtypes;
* ECOG 0~1;
* Major organ function is normal (14 days prior to enrollment) if the following criteria are met:

  1. The blood routine examination criteria should meet (no blood transfusion and no granulocyte colony stimulation agent treatment within 14 days before enrollment): HB≥90 g/L; ANC≥1.5×109 /L; PLT≥100×109 /L;
  2. Non-functional organic diseases shall meet the following criteria: T-BIL≤1.5×ULN (upper limit of normal value); ALT and AST≤2.5 x ULN; Serum creatinine ≤2×ULN, or endogenous creatinine clearance ≥ 30ml/min(Cockcroft-Gault formula);
* Subjects (or their legal representatives) must sign an informed consent form (ICF) indicating that they understand the purpose and procedures of the study and are willing to participate in the study.
* Pregnant women must have a negative pregnancy test result (beta-hCG) (urine or serum) within 7 days before the first administration of the randomized or study drug.

Exclusion Criteria:

* Histopathological examination revealed any small cell component of ureter or pelvis, simple adenocarcinoma, simple squamous cell carcinoma, or simple squamous CIS;
* Previous treatment with other PD-1/PD-L1 inhibitors and/or HER-2 inhibitors;
* Active malignancies other than the disease being studied for treatment (i.e., disease progression within the last 24 months or requiring a change in treatment), only the following special cases are allowed: i. Skin cancer that has been treated within the last 24 months and has been completely cured ii. Adequately treated lobular carcinoma in situ (LCIS) and ductus CIS iii. History of local breast cancer and is receiving antihormonal drugs or history of local prostate cancer (N0M0) and is receiving androgen blocking therapy;
* History of uncontrolled cardiovascular disease, including: 1) any of the following in the past 3 months: unstable angina pectoris, myocardial infarction, ventricular fibrillation, torsion ventricular tachycardia, cardiac arrest, or known congestive New York Heart Association Class III-IV heart failure, cerebrovascular accident, or transient ischemic attack; 2) QTc interval prolongation confirmed by ECG evaluation at screening (Fridericia; QTc > 480 ms); 3) Pulmonary embolism or other venous thromboembolism within the past 2 months;
* Pregnant or lactating women;
* Human immunodeficiency virus (HIV) infection is known unless the subject has been on stable antiretroviral therapy for the past 6 months or longer, has not developed an opportunistic infection in the past 6 months, and has a CD4 count > 350 in the past 6 months.
* Known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., HBV DNA positive (>1×104 copies /mL or >2000 IU/ml) must be excluded for known hepatitis B virus (HBV) carriers; Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis];
* Have not recovered from the toxic effects of previous anticancer treatment (except for those that are not clinically significant, such as hair loss, skin discoloration, neuropathy, and hearing impairment);
* Delayed wound healing, defined as skin/bedsore ulcers, chronic leg ulcers, known stomach ulcers, or non-healing of incisions;
* Major surgery within 4 weeks before day 1 of Cycle 1 (TURBT is not considered a major surgery);
* Other patients assessed by the investigator as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Kidney-intact disease-free survival, KI-DFS | Up to 12 months
  Defined as the time to systemic relapse or death.

SECONDARY OUTCOMES:
Time to progression, TTP | Up to 3 years
  Defined as the time to systemic progression or death.
Time to RNU | Up to 3 years
  Defined by time from day of first treatment to RNU.
Disease-specific survival time, DSS | Up to 3 years
  Defined by time from day of first treatment to death due to a specific disease, reflecting the clinical benefit of a specific disease.
Overall survival | Up to 3 years
  Defined by time from day of first treatment to death.
3m complete remission | Up to 3 years
  CR is defined by CT urography

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No